# Efficacy of mirabegron for treatment of nocturnal enuresis in children

## Introduction

Enuresis is an extremely common condition, which, although somatically benign, poses long-term psychosocial risks if untreated.

Nocturnal enuresis (NE) or bedwetting is defined as the voluntary or involuntary wetting of clothes or bedding with urine for a period of at least 3 consecutive months in children older than 5 years of age. It affects 15% - 20% of children aged 5 years, and 1% - 2% of adolescents[2]. Although spontaneous recovery occurs at a rate of 10–15% per year[3], NE still has a certain impact on the child's social, emotional and psychological development. According to the International Children's Continence Society (ICCS) recommendation, NE can be subclassified into monosymptomatic nocturnal enuresis (MNE) and non-monosymptomatic nocturnal enuresis (NMNE) based on whether accompanied with lower urinary tract symptoms (LUTS) or not[4]. MNE is defined as involuntary urine voiding during sleep without other LUTS, such as daytime urinary frequency, urgency, or incontinence of urine. More than 68.5% of NE patients are MNE[5].

Various interventions including pharmacological, behavioral and other approaches have been used for the treatment of MNE. Alarm therapy, one of the first line treatment, has been proved to be effective for MNE and should be first taken into consideration in children under 8 year age with adequate family support[6]. Desmopressin is the most widely used medical treatment in the management of MNE[7]. Combine therapy of desmopressin plus anticholinergics is often taken

into consideration when the patients are refractory to single treatment, having behavioral problems or frequent nighttime enuresis[8].

## Aim

To evaluate the efficacy of B3 agonist mirabegron in the management of nocturnal enuresis in children.

# **Patients & Methods:**

The study will be conducted in urology department, Menoufia University Hospital.

Sample size: 151

#### **Inclusion criteria:**

Children from 5-15 years old

Nocturnal enuresis

#### **Exclusion criteria:**

Patients with anatomical lower urinary tract abnormalities

Any neurological diseases

Experienced treatment failure

Active urinary tract infection

#### **Preintervention assessment:**

## Laboratory investigations:

Urine analysis and urine culture & sensitivity

## **Radiological investigation:**

Ultrasound abdomen and pelvis

The main outcomes included complete response rate, success rate, mean number of wet nights per week at the end of treatment, relapse rate at the end of following up, and adverse events during the treatment. According to the definition of ICCS, the outcomes were evaluated as follows: (1) complete response (CR) as a 100 % decrease; (2) response (R) as a ≥90 % decrease; (3) partial response (PR) as a 50–89 % decrease; (4) non-response (NR) as 0–49 % decrease in the number of wet nights. Relapse was defined as reappearance of >1 wet night per week for complete responders or >50% of pretreatment wetting frequency for partial responders. CR, R, and PR were regarded as the success.

## **Results:**

The results will be recorded, tabulated, and statistically analyzed.

## **Discussion:**

The results will be discussed in comparison to those mentioned in the literature.

# **References:**

- 1. Neveus T, von Gontard A, Hoebeke P, Hjalmas K, Bauer S, Bower W, et al. The standardization of terminology of lower urinary tract function in children and adolescents: report from the Standardisation Committee of the International Children's Continence Society. The Journal of urology. 2006;176(1):314-24.
- 2. Neveus T. Nocturnal enuresis-theoretic background and practical guidelines. Pediatric nephrology (Berlin, Germany). 2011;26(8):1207-14.

- 3. Cakiroglu B, Tas T, Eyyupoglu SE, Hazar AI, Can Balci MB, Nas Y, et al. The adverse influence of spina bifida occulta on the medical treatment outcome of primary monosymptomatic nocturnal enuresis. Archivio italiano di urologia, andrologia : organo ufficiale [di] Societa italiana di ecografia urologica e nefrologica.2014;86(4):270-3.
- 4. Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, et al. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourology and urodynamics. 2016;35(4):471-81.
- 5. Franco I, von Gontard A, De Gennaro M, International Childrens's Continence S. Evaluation and treatment of nonmonosymptomatic nocturnal enuresis: a standardization document from the International Children's Continence Society. Journal of pediatric urology. 2013;9(2):234-43.
- Van Leerdam FJ, Blankespoor MN, Van Der Heijden AJ, Hirasing RA. Alarm treatment is successful in children with day- and night-time wetting.
  Scandinavian journal of urology and nephrology. 2004;38(3):211-5. doi: 10.1080/00365590410025460. PubMed PMID: 15204373.
- 7. Alloussi SH, Wuertz G, Lang C, Madersbacher H, Strugala G, Seibold J, et al. Desmopressin treatment regimens in monosymptomatic and nonmonosymptomatic enuresis: A review from a clinical perspective. Journal of pediatric urology. 2011;7(1):10-20. PubMed PMID: WOS:000291195600003.
- 8. Leebeek-Groenewegen A, Blom J, Sukhai R, Van Der Heijden B. Efficacy of desmopressin combined with alarm therapy for monosymptomatic nocturnal enuresis. The Journal of urology. 2001;166(6):2456-8. PubMed PMID: 11696811.